CLINICAL TRIAL: NCT01866384
Title: Safety and Tolerability of a Protocol of Targeted Temperature Management After Intracerebral Hemorrhage
Brief Title: Targeted Temperature Management After Intracerebral Hemorrhage
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 12D.466
Record Dates: First submitted 2013-05-20; First posted 2013-05-31 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Cerebral Hemorrhage; Hypothermia
MeSH Terms: conditions — Cerebral Hemorrhage; Hypothermia | interventions — Hypothermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Temperature (Other): 72 hours of Normal Temperature (36-37 degrees Celcius). Subjects in all arms will otherwise receive identical therapeutic interventions pre-defined by our local IPH management protocol.
  Interventions: Other: Normal Temperature
- Mild Induced Hypothermia (Experimental): 72 hours of mild induced hypothermia (32-34 degrees Celcius). Subjects in all arms will otherwise receive identical therapeutic interventions pre-defined by our local IPH management protocol.
  Interventions: Procedure: mild induced hypothermia

INTERVENTIONS:
Procedure: mild induced hypothermia — Patients with intraparancymal hemorrhage within 6 hours of onset will be randomized to either the mild induced hypothermia group or the normal temperature group (control). In this arm, the patient will have 72 hours of Targeted Temperature Managment to mild induced hypothermia (32-34 degrees Celcius).
  Arms: Mild Induced Hypothermia
Other: Normal Temperature — In this arm, the patient will have standard of care intraparenchymal hemorrhage management per institutional policy, with normal body temperature management (36-37 degrees Celcius).
  Arms: Normal Temperature

SUMMARY:
Early hematoma growth (HG) after spontaneous intra-cerebral/intra-parenchymal hemorrhage (IPH) is common and associated with neurological deterioration and poor clinical outcome. Temperature modulation to hypothermia (Temperature, 32-34°C) has been associated with reduction or improvement of physiopathologic processes associated with inflammatory activation and degradation of blood-brain barrier after all types of brain injury. In this sense, we believe that the initiation of an ultra-early protocol of active temperature modulation or Targeted Temperature Management (TTM) to mild induced hypothermia (MIH, 32-34°C) may be associated with good safety and tolerability profile, less HG and cerebral edema after IPH by modulation of systemic and local inflammatory responses, so we hypothesize that TTM to MIH will be a safe/tolerable and effective therapy to limit HG and cerebral edema after IPH.

DETAILED DESCRIPTION:
In this randomized clinical trial, patients with IPH within 6 hours of onset will be randomized to one of two study arms. In one arm, patients will have 72 hours of TTM to MIH (32-34 degree Celcius). In the second arm, patients will have 72 hours of TTM to Normal Temperature (NT)(36-37 degrees Celcius). Subjects in all arms will otherwise receive identical therapeutic interventions pre-defined by our local IPH management protocol.

Primary outcomes are examining the frequency of adverse events (AEs) that will be possibly or probably related to treatment. AEs will be assessed up to 15-days after admission or discharge if earlier and the frequency of severe adverse events (SAEs) that will be possibly and probably related to treatment.

SAEs will be assessed up to 90-days.

The secondary outcome measures will be in-hospital neurological deterioration between day 0-7 (decrease in GCS10 in ≥2 points, or increase in the NIHSS11 ≥4 points), in-hospital mortality, modified Rankin Score [mRS]12 at discharge and 90-days.

To determine whether TTM to MIH can limit HG and cerebral edema, will be examining absolute change in hematoma between baseline and 24 hours, new or absolute change in IVH between baseline and 24 hours, the proportion of patients with HG, absolute change in hemostatic proteins, the absolute change in cerebral edema between baseline and 24, 48,72, and 168-hours, relative change in cerebral edema.

ELIGIBILITY:
Inclusion Criteria:

* spontaneous supratentorial IPH documented by CT scan within 6 hours after the onset of symptoms and admission to the Neuro-ICU,
* baseline hematoma >15cc with or without IVH
* need for mechanical ventilation

Exclusion Criteria:

* GCS <6
* age <18 years
* pregnancy
* pre-morbid mRS>2
* Do Not Resuscitate (DNR) order "prior" to enrollment
* uncontrolled bleeding of different etiology (trauma, gastro-intestinal bleeding [UGIB/LGIB]
* planned surgical decompression within 24 hours
* secondary causes of IPH (ischemic stroke, coagulopathy [INR>1.4, aPTT> 1.5 times baseline, thrombocytopenia platelets <100,000/uL], trauma, AVM, aneurysm, cerebral sinus thrombosis, or other causes)
* evidence of sepsis
* inability to obtain written informed consent
* participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) that will be possibly or probably related to the treatment. | Continuous throughout 3 year study period
  To determine whether TTM to MIH is safe and tolerable after IPH measured by the frequency of adverse events (AEs) that will be possibly or probably related to the treatment.

SECONDARY OUTCOMES:
In-hospital neurological deterioration between day 0-7. | Continuous throughout 3 year study period
  To determine whether TTM to MIH can limit hematoma growth and cerebral edema measured by in-hospital neurological deterioration between day 0-7.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Rincon, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States